CLINICAL TRIAL: NCT00289120
Title: Effect of Cola on Urinary Stone Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kenneth Ogan, MD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 0133-2003; GCRC#2403
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Stone
Keywords: urolithiasis, cola
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cola beverage (Experimental): Subjects will be given 500cc of Cola twice daily.
  Interventions: Drug: Cola beverage
- Deionized water (Placebo Comparator): Subjects will be given 500cc of deionized water.
  Interventions: Drug: Deionized water

INTERVENTIONS:
Drug: Cola beverage — Subjects will be given 500cc of Cola beverage twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.There will be a three weeks interval before crossover to the other treatment arm.
  Arms: Cola beverage
Drug: Deionized water — Subjects will be given 500cc of deionized water to be ingested twice daily with breakfast and dinner for three weeks while on a metabolic diet. There will be a three weeks interval before crossover to the other treatment arm
  Arms: Deionized water

SUMMARY:
Examine the effects of cola on risks of kidney stones

DETAILED DESCRIPTION:
Prospective crossover study examining the risks of cola on stone risk factors.

ELIGIBILITY:
Inclusion Criteria:

* urolithiasis, healthy volunteer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Herrel L, Pattaras J, Solomon T, Ogan K. Urinary stone risk and cola consumption. Urology. 2012 Nov;80(5):990-4. doi: 10.1016/j.urology.2012.07.003. Epub 2012 Sep 25. PMID 23017784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited patients of Emory University Department of Urology
Pre-assignment Details: Normal subjects and calcium oxalate stone-formers were included.
Groups:
- Cola First, Then Water: Phase 1: Subjects will be given 500cc of Cola beverage twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.
  There will be a three weeks wash-out period before patients entere phase 2 of thre study.
  Phase 2: Subjects will be given 500cc of deionized water twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.
Period: Overall Study
Arm/Group | Cola First, Then Water
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Thirteen subjects, including 10 normal subjects and 3 calcium oxalate stone-formers were enrolled in this prospective cross-over study.
Groups:
- Cola First, Then Water: Phase 1: Subjects will be given 500cc of Cola beverage twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.
  There will be a 3-week wash out period before subjects enter phase 2 of the study.
  Phase 2: Subjects will be given 500 cc of deionized water beverage twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.
Arm/Group | Cola First, Then Water
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Study participants [Number; unit: participants]
  Normal subjects | 10
  Calcium oxalate stone- formers | 3

OUTCOME MEASURES:

1. Primary Outcome: The Plasma and Urine Parameters
Description: The Plasma and Urine Parameters that were assessed at the end of cola and water (arms) phase:
  Plasma Parameters:
  CA (mg per dL) GLU (mg per dL) BUN (mg per dL) Cr (mg per dL) Prot (mg per dL) ALB (mg per dL)
  Urine Parameters:
  uCa (mg per dL) uMg (mg per dL) uP (mg per dL) uCr (mg per dL) uCit (mg per dL) uOx (mg per dL) uUA (mg per dL)
  The parameters were consolidated into the one value as a mean of all the values in the phase or group (Table 3) and later for longitudinal analysis as a mean of all the values in the phase for each participant (Table 4).
  measure of dispersion was standard deviation.
Time Frame: at the end of each 6-day intervention in Cola and Water Phase
Measure: Mean (Standard Deviation); unit: mg per dL
Groups:
- Cola: they ingested 500 mL of cola (regular Publix brand©) twice daily, with breakfast and dinner.
- Water: participants ingested 500 mL of deionized water twice daily, with breakfast and dinner.
Arm/Group | Cola | Water
Number analyzed (Participants) | 13 | 13
mg per dL
  Plasma Proteins | 6800 (500) | 6800 (500)
  Plasma Albumin | 3700 (300) | 3700 (300)
  Plasma Calcium | 9.1 (0.3) | 9.0 (0.2)
  Mean Plasma Glucose | 92.8 (9) | 95.2 (15.7)
  blood urea nitrogen | 10.1 (4.5) | 11.1 (5.0)
  Plasma Creatinine | 0.9 (0.2) | 2.1 (2.9)
  Urinary Calcium | 124.3 (74.5) | 146.4 (86.9)
  Urinary Magnesium | 94.6 (43.7) | 106.8 (49.9)
  Urinary Phosphets | 720.7 (224.1) | 739.6 (320.5)
  Urinary Creatinine | 1620.1 (699.0) | 1950.1 (1057.1)
  Urinary Citrate | 475.9 (240.6) | 727.7 (666.2)
  Urinary Oxalates | 39.7 (25.6) | 34.7 (21.0)
  Uric acids | 555.3 (183.1) | 646.4 (272.0)

2. Primary Outcome: The Plasma and Urine Parameters
Description: The Plasma and Urine Parameters that were assessed at the end of cola and water (arms) phase:
  Plasma Parameters:
  Na (mEq per L) K (mEq per L) CL (mEq per L) CO2(mEq per L) AG (mEq per L)
  The parameters were consolidated into the one value as a mean of all the values in the phase or group (Table 3) and later for longitudinal analysis as a mean of all the values in the phase for each participant (Table 4).
  measure of dispersion was standard deviation.
Time Frame: at the end of 6-day intervention of Cola and water phase
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Water | Cola
Number analyzed (Participants) | 13 | 13
mEq/L
  Plasma sodium | 138.3 (2.5) | 139.1 (2.3)
  Plasma Potassium | 3.8 (0.2) | 3.9 (0.4)
  Plasma Chlorides | 104.8 (2.3) | 105.2 (3.0)
  Plasma CO2 | 26.1 (2.0) | 26.4 (2.4)
  Plasma AG | 7.3 (1.2) | 7.3 (1.6)

3. Primary Outcome: The Plasma Osmolarity
Description: The Plasma osmolarity that were assessed at the end of cola and water (arms) phase:
  Plasma Parameters:
  OSM (mOsm/L)
  The parameters were consolidated into the one value as a mean of all the values in the phase or group (Table 3) and later for longitudinal analysis as a mean of all the values in the phase for each participant (Table 4).
  measure of dispersion was standard deviation.
Time Frame: at the end of 6-day intervention of cola and water phase
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Water | Cola
Number analyzed (Participants) | 13 | 13
mOsm/L | 276.5 (4.8) | 277.5 (5.0)

4. Secondary Outcome: Total Urine Volume
Description: The Plasma and Urine Parameters that were assessed at the end of cola and water (arms) phase:
  Urine Parameters:
  Total Urine Volume (mL/day)
  The parameters were consolidated into the one value as a mean of all the values in the phase or group (Table 3) and later for longitudinal analysis as a mean of all the values in the phase for each participant (Table 4).
  measure of dispersion was standard deviation.
Time Frame: at the end of each 6-day intervention in Cola and Water Phase
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Water | Cola
Number analyzed (Participants) | 13 | 13
mL/day | 2521.3 (1152.6) | 2266.2 (811.0)

5. Secondary Outcome: Urinary pH
Description: The Urine pH that were assessed at the end of cola and water (arms) phase The parameters were consolidated into the one value as a mean of all the values in the phase or group (Table 3) and later for longitudinal analysis as a mean of all the values in the phase for each participant (Table 4).
  measure of dispersion was standard deviation.
Time Frame: at the end of each 6-day intervention in Cola and Water Phase
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cola | Water
Number analyzed (Participants) | 13 | 13
pH | 6.0 (0.6) | 6.0 (0.5)

6. Primary Outcome: The Plasma and Urine Parameters
Description: The Urine Parameters that were assessed at the end of cola and water (arms) phase:
  Urine Parameters:
  uNa (mEq per d) uK (mEq per d)
  The parameters were consolidated into the one value as a mean of all the values in the phase or group (Table 3) and later for longitudinal analysis as a mean of all the values in the phase for each participant (Table 4).
  measure of dispersion was standard deviation.
Time Frame: at the end of 6-day intervention of Cola and water phase
Measure: Mean (Standard Deviation); unit: mEq per d
Arm/Group | Water | Cola
Number analyzed (Participants) | 13 | 13
mEq per d
  Urinary sodium | 139.9 (40.0) | 103.9 (43.5)
  Urinary Potassium | 49.3 (31.4) | 41.4 (17.1)

ADVERSE EVENTS:
Groups:
- Cola Beverage Phase: Subjects were given 500cc of Cola twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.
  There will be a three weeks interval (wash out period) before crossover to the other treatment arm.
  No adverse event reported.
- Deionized Water Drinking Phase: Subjects were given 500cc of regular deionized water twice daily to be ingested with breakfast and dinner for six days while on a metabolic diet.
  No adverse event reported.
Arm/Group | Cola Beverage Phase | Deionized Water Drinking Phase
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No